#### STATISTICAL ANALYSIS PLAN

A Multicenter, Randomized, Double-blind, Vehicle-controlled, Parallel-group Comparison Trial to Demonstrate the Superiority of 1% OPA-15406 Ointment to the Vehicle in Adult Patients with Atopic Dermatitis (Phase 3 Trial)

NCT Number: 03908970

PRT NO.: 271-102-00007

Version Date: 25 February 2020 (Version 1.0)

#### Otsuka Pharmaceutical Co., Ltd.

#### Investigational Medicinal Product OPA-15406

Protocol No. 271-102-00007

A Multicenter, Randomized, Double-blind, Vehicle-controlled, Parallel-group Comparison Trial to Demonstrate the Superiority of 1% OPA-15406 Ointment to the Vehicle in Adult Patients with Atopic Dermatitis (Phase 3 Trial)

Statistical Analysis Plan

Version: 1.0
Issue Date: 25 Feb 2020
Clinical Protocol Version 3.0 Date: 25 Feb 2019

## Confidential

May not be used, divulged, published, or otherwise disclosed without the prior written consent of Otsuka Pharmaceutical Co., Ltd.

## **Table of Contents**

| Tabl | Table of Contents 2 | |
|-------|------------------------------------------|----|
| List | of Appendices | 4 |
| List | of Abbreviations and Definition of Terms | 5 |
| 1 | Introduction | 6 |
| 2 | Trial Objectives | 6 |
| 3 | Trial Design | 6 |
| 3.1 | Type/Design of Trial | 6 |
| 3.2 | Methods of Administration | 7 |
| 3.2.1 | Dose, Regimen, and Treatment Period | 7 |
| 3.2.2 | Treatment Area | 8 |
| 3.3 | Trial Population | 8 |
| 3.4 | Trial Visit Window | 9 |
| 4 | Sample Size | 10 |
| 5 | Statistical Analysis Datasets | 10 |
| 5.1 | Full Analysis Set (FAS) | 10 |
| 5.2 | Safety Set (SS) | 10 |
| 5.3 | Handling of Missing Data | 11 |
| 6 | Primary and Secondary Outcome Variables | 11 |
| 6.1 | Primary Outcome Variable | 11 |
| 6.2 | Secondary Outcome Variables | 11 |
| 7 | Disposition and Demographic Analysis | 11 |
| 7.1 | Subject Disposition | 11 |
| 7.2 | Demographic and Baseline Characteristics | 12 |
| 7.3 | Baseline Disease Evaluation | 12 |
| 7.4 | Treatment Compliance | 12 |
| 7.5 | Prior and Concomitant Medications | 13 |
| 7.6 | Protocol Deviations | 13 |
| 8 | Efficacy Analysis | 13 |
| 8.1 | Primary Efficacy Endpoint | 13 |
| 8.1.1 | Primary Efficacy Analysis | 13 |

| 8.2 | Secondary Efficacy Endpoints | 14 |
|---|---|---|
| 8.2.1 | Success Rates in IGA (Revised Definition) and EASI | 14 |
| 8.2.2 | Change From Baseline Through Week 4 in the IGA Score | 14 |
| 8.2.3 | Shift Table for Investigator's Global Assessment Scores up to Week 4 | 16 |
| 8.2.4 | Change From Baseline Through Week 4 in the Total EASI Score and Each EASI Clinical Sign Score | 16 |
| 8.2.5 | Change From Baseline Through Day 8 in VRS for Pruritus | 16 |
| 8.2.6 | Change From Baseline Through Week 4 in VRS for Pruritus | 16 |
| 8.2.7 | Change From Baseline Through Week 4 in the Total POEM Score | 16 |
| 8.2.8 | Change From Baseline Through Week 4 in Skindex-16 | 16 |
| 8.2.9 | Change From Baseline Through Week 4 in the Total Affected BSA (%) | 17 |
| 8.3 | Subgroup Analyses | 17 |
| 9 | Safety Analysis | 17 |
| 9.1 | Extent of Exposure | 17 |
| 9.2 | Adverse Events | 17 |
| 9.3 | Clinical Laboratory Tests | 18 |
| 9.4 | Vital Signs and Body Weight | 18 |
| 9.5 | Physical Examination | 19 |
| 9.6 | Electrocardiogram | 19 |
| 9.7 | Liver Function Tests | 19 |
| 10 | Pharmacokinetic Analysis | 19 |
| 11 | Pharmacodynamic Analysis | 19 |
| 12 | Pharmacogenomic Analysis | 19 |
| 13 | Interim Analysis | 19 |
| 14 | Changes in the Planned Analyses | 19 |
| 15 | References | 20 |

## **List of Appendices**

| Appendix 1 | Criteria for Vital Signs Potential Clinical Significance | 21 |
|------------|----------------------------------------------------------|----|
| Appendix 2 | Criteria for Potential Hy's Law | 22 |
| Appendix 3 | List of Summary Tables | 23 |
| Appendix 4 | List of Subject Data Listings | 36 |

## **List of Abbreviations and Definition of Terms**

#### **List of Abbreviations**

| <b>Abbreviation</b> | Expansion or Definition |
|---------------------|----------------------------------------------|
| AE | Adverse event |
| BMI | Body mass index |
| BSA | Body surface area |
| CRF | Case report form |
| EASI | Eczema Area and Severity Index |
| FAS | Full Analysis Set |
| IGA | Investigator's Global Assessment |
| IMP | Investigational medicinal product |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed Model Repeated Measures |
| OC | Observed Cases |
| POEM | Patient-Oriented Eczema Measure |
| SS | Safety Set |
| TEAE | Treatment-emergent adverse event |
| VRS | Verbal Rating Scale |

### **List of Definitions of Terms**

| <u>Term</u> | <u>Definition</u> |
|---|---|
| Descriptive statistics | Number of subjects, mean, standard deviation, maximum, |
| | median, and minimum |
| Frequency distribution | Number and percentage of subjects |

#### 1 Introduction

This statistical analysis plan describes in detail the methodology for statistical analysis planned in the protocol for Trial 271-102-00007.

## 2 Trial Objectives

Primary Objective: To demonstrate the superiority of 1% OPA-15406 ointment to the vehicle when administered the investigational medicinal product (IMP; 1% OPA-15406 ointment or vehicle) twice daily for 4 weeks in adult patients with atopic dermatitis (AD), using success rate in Investigator's Global Assessment (IGA) at Week 4 as the primary endpoint.

Secondary Objective: To evaluate the efficacy (secondary endpoint) and safety of 1% OPA-15406 ointment when administered the IMP twice daily for 4 weeks in adult patients with AD.

## 3 Trial Design

#### 3.1 Type/Design of Trial

This trial is a multicenter, randomized, double-blind, vehicle-controlled, parallel-group comparison trial to demonstrate the superiority of 1% OPA-15406 ointment to the vehicle in adult AD patients. This trial consists of the 1% OPA-15406 group and the vehicle group. The trial design is shown in Figure 3.1-1.

#### 1) Screening period

After obtaining informed consent, the investigator or subinvestigator will perform a screening examination. The screening period is defined as the period between the day of screening examination and the day of baseline examination (2 to 30 days).

#### 2) Assessment period (treatment period)

The assessment period is defined as the period between the day of baseline examination and the end of Week 4 examination (or the end of withdrawal examination). The subjects who meet the inclusion and exclusion criteria at the baseline examination will be allocated to 1% OPA-15406 ointment or the comparator (vehicle [placebo]). The allocated IMP will be administered to the treatment area from the day of the baseline examination twice daily for 4 weeks. After the baseline examination, the examinations will be performed at Weeks 1, 2, and 4.

If a subject discontinues the IMP administration between the day of the baseline examination and the day of the Week 4 examination, a withdrawal examination will be performed for that subject.

#### 3) Trial period

The trial period for individual subjects is the period from the day of obtaining the subject's written informed consent to the day of the Week 4 examination or withdrawal examination. For subjects who missed the Week 4 examination or withdrawal examination, the day of discontinuation will be the day when the investigator or subinvestigator determined that the subject was to be withdrawn from the trial. It does not include the follow-up period for adverse events (AEs).



Figure 3.1-1 Trial Design

#### 3.2 Methods of Administration

#### 3.2.1 Dose, Regimen, and Treatment Period

The 1% formulation or the vehicle of OPA-15406 ointment will be administered twice daily (approximately 12 hours apart between morning and night administration) for 4 weeks. The amount of IMP (g) per dose is  $10 \text{ g/m}^2$  BSA and calculated as follows.

1) The subject's BSA (m<sup>2</sup>) will be calculated based on height and body weight at the screening examination, using the following equation.

BSA (m<sup>2</sup>) = 
$$\sqrt{\frac{\text{Ht (cm)} \times \text{Wt (kg)}}{3600}}$$

BSA = body surface area; Ht = height; Wt: body weight (Mosteller 1987)

- 2) The treatment area will be specified.
- 3) The amount of IMP (g) per dose will be calculated as "subject's BSA (m²)" × "treatment area (%)" × "10 g/m²."

  Example: In case of a BSA of 0.7m² and an affected BSA of 32%: 0.7 m² × 0.32 × 10 g/m² = 2.24g

#### 3.2.2 Treatment Area

The treatment area with the IMP is defined as follows.

- The treatment area selected at the baseline examination will be the affected area determined at the baseline examination.
- After the baseline examination, when the affected area has expanded or a new affected area is detected, the expanded or newly affected area will also be included in the treatment area.
- Even when the affected area is relieved, the IMP administration should be continued there as the treatment area.

The investigator or subinvestigator will instruct the subject regarding the method of administration by specifying the treatment area (%) and the total amount of administration (g) for each treatment area using the human body drawing, and will give the human body drawing (copy) to the subject. The investigator or subinvestigator will record the treatment area (%) of the 4 body regions (face, neck, and head [excluding scalp]; upper limbs; trunk; and lower limbs) in the source document and case report form (CRF).

#### 3.3 Trial Population

The target population of this trial is adult AD patients with an IGA score of 2 or 3. Subjects will be included in the trial to reach the target number of 340 subjects for IMP administration. Any withdrawal will not be supplemented.

#### 3.4 Trial Visit Window

The start date of IMP administration is defined as baseline (Day 1) to count the number of days after starting IMP administration. Unscheduled visit data and withdrawal visit data as well as scheduled visit data will be included to determine timepoints for analysis. For efficacy endpoints, data up to 3 days after the end of IMP administration (final day of IMP administration + 3 days) will be included in the analysis. For safety endpoints, all data from the first IMP administration will be included in the analysis. Timepoints for analysis and acceptable windows are shown in Table 3.4-1. If there are multiple data points within an acceptable window, the last one in the window will be used. The Last Visit data for efficacy endpoints will be from the last visit during the period from the day after the first day of IMP administration (Day 2) through the third day after the last IMP administration (including unscheduled and withdrawal visit data), and those for safety endpoints will be from the last visit available from all data after the first day of IMP administration.

The baseline data for analysis will be from the visit closest and prior to the first day of IMP administration.

For the Verbal Rating Scale (VRS), the patient diary will be used as the source of data for the period from the start date of IMP administration (Day 1) through Day 8. After Week 1, CRF Visit data (including unscheduled and withdrawal visit data) excluding patient diary data will be used to specify the timepoints for analysis according to Table 3.4-1. If there are multiple data points within an acceptable window, the last one in the window will be used.

| Table 3.4-1 Timepoints and Acceptable Windows for Efficacy and Safety Endpoints | | | | |
|---|---|---|---|---|
| Timepoint | Target Day | Interval (day | s after starting adı | ministration) |
| Baseline | 1 | _ | to | 1 |
| 1 day after start of IMP<br>administration (VRS alone) | 2 | _ | to | _ |
| 2 days after start of IMP<br>administration (VRS alone) | 3 | _ | to | _ |
| 3 days after start of IMP administration (VRS alone) | 4 | _ | to | _ |
| 4 days after start of IMP administration (VRS alone) | 5 | _ | to | _ |
| 5 days after start of IMP administration (VRS alone) | 6 | _ | to | _ |
| 6 days after start of IMP administration (VRS alone) | 7 | _ | to | _ |
| 7 days after start of IMP administration (VRS alone) | 8 | _ | to | _ |
| 8 days after start of IMP administration (VRS alone) | 9 | _ | to | _ |
| Week 1 | 8 | 2 | to | 10 |
| Week 2 | 15 | 11 | to | 21 |
| Week 4 | 29 | 22 | to | 32 |

## 4 Sample Size

In the phase 2 trial in adult patients in Japan (Trial 271-15-001), the success rate in IGA was 22.4% and 9.1% in the 1% OPA-15406 group and the vehicle group, respectively. With the assumption that a similar success rate is obtained in each group, 167 subjects are necessary to achieve a power of 90% at a two-sided significance level of 5%. Therefore, the target sample size is 170 subjects in each group, a total of 340 subjects.

## 5 Statistical Analysis Datasets

## 5.1 Full Analysis Set (FAS)

The FAS consists of all subjects who have received the IMP at least once.

## 5.2 Safety Set (SS)

The SS consists of all subjects who have received the IMP at least once.

#### 5.3 Handling of Missing Data

For the success rate in IGA, the primary endpoint, subjects with missing IGA data will be handled as non-responders. Subjects with only baseline values or with data missing at any timepoint will also be handled as non-responders.

## 6 Primary and Secondary Outcome Variables

#### 6.1 Primary Outcome Variable

Success rate in IGA at Week 4: percentage of subjects with IGA score of 0 or 1 with improvement by at least 2 grades.

#### 6.2 Secondary Outcome Variables

- Success rate in IGA at Week 4: percentage of subjects with improved IGA score of 0 or 1 (revised definition from primary outcome variable)
- Change from baseline at Week 4 in the IGA score
- Success rate in EASI 75 (improvement of ≥75% in EASI), EASI 90 (improvement of ≥90% in EASI), and EASI 50 (improvement of ≥50% in EASI) at Week 4
- Change from baseline at Week 4 in the total EASI score and each EASI clinical sign score
- Change from baseline at Week 4 in VRS for pruritus
- Change from baseline through Day 8 in VRS for pruritus
- Change from baseline at Week 4 in the total Patient-Oriented Eczema Measure (POEM) score
- Change from baseline at Week 4 in each item score, the scale score (mean score of item scores on each scale [symptoms, emotions, and functions]), and the mean score of 16 items of Skindex-16
- Change from baseline at Week 4 in the total affected BSA (%)

## 7 Disposition and Demographic Analysis

#### 7.1 Subject Disposition

The number of subjects screened and the number of subjects allocated will be calculated. Unless specified otherwise, the following tabulations will be presented by treatment group (1% OPA-15406 or vehicle). Frequency distribution (number and percentage, the same hereinafter) will be provided for subjects who received, who completed, and who discontinued IMP administration. Also, the number and percentage of subjects included

in the statistical analysis datasets will be presented. The number of allocated subjects will be used as the denominator to calculate the percentage. For subjects who discontinued treatment, the frequency distribution by reason for discontinuation will be presented.

#### 7.2 Demographic and Baseline Characteristics

Based on the FAS and SS, age, sex, disease duration, body weight, height, body mass index (BMI), race, and severity of AD will be presented by treatment group and in total. The descriptive statistics will be presented for age, disease duration, body weight, height, and BMI; and frequency distribution for sex, race, and severity of AD. Medical histories and complications will be coded by System Organ Class (SOC) and Preferred Term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA). Medical histories and complications will be listed but not summarized.

For the computation of disease duration, date data that are partially missing will not be imputed. Where the month and day are missing, only the year will be used, and where the day is missing, the year and month will be used for calculation.

```
Where the "year, month, and day" are available:
(Year-Month-Day – Year-Month-Day + 1) / 365.25
```

Where only the "year and month" are available:

$$[(Year \times 12 + Month) - (Year \times 12 + Month) + 1] / 12$$

Where only the "year" is available: Year - Year + 1

#### 7.3 Baseline Disease Evaluation

Based on the FAS and SS, the frequency distribution of baseline IGA scores (2 or 3) and the descriptive statistics for the total EASI (Eczema Area and Severity Index) score at baseline will be presented by treatment group and in total. The affected area at baseline will be classified in the following categories, and the frequency distribution calculated by treatment group and in total.

Affected area categories:  $\geq 5\%$  to  $\leq 10\%$ ,  $\geq 10\%$  to  $\leq 30\%$ , and  $\geq 30\%$ 

#### 7.4 Treatment Compliance

Based on the SS, the compliance with the amount and number of doses from the baseline through Week 4 will be classified in the following categories, and the number and percentage of subjects will be calculated by treatment group and for all subjects. Also, the number and percentage of subjects administered will be calculated by week (Weeks 1, 2, 3, 4, 5, and Any Exposure). The method for calculating compliance will be defined in a separate analysis data set specification, etc.

Categories for compliance with the amount and number of doses:

<50%,  $\ge 50\%$  to <60%,  $\ge 60\%$  to <70%,  $\ge 70\%$  to <80%,  $\ge 80\%$  to <90%,  $\ge 90\%$  to <100%,  $\ge 100\%$  to <110%,  $\ge 110\%$  to <120%, and  $\ge 120\%$ 

Where the weight of IMP at retrieval is unknown, the amount of administration will be calculated by assuming that the retrieved weight is 0.

#### 7.5 Prior and Concomitant Medications

Based on the SS, the number and percentage of subjects taking medications before the start of, during, and after the end of IMP administration will be calculated for each medication by treatment group and in total. Medications will be coded using WHO Drug Dictionary and summarized by ATC classifications level 2 and preferred name. Concomitant therapies will be listed but not summarized.

#### 7.6 Protocol Deviations

Based on the allocated subjects, the number and percentage of subjects with major protocol deviations will be presented by treatment group and in total. Also for each site, the number and percentage of subjects with major protocol deviations will be presented by treatment group and in total.

## 8 Efficacy Analysis

Based on the FAS, the following analysis will be performed.

#### 8.1 Primary Efficacy Endpoint

The primary endpoint is the success rate in IGA at Week 4 (percentage of subjects with IGA score of 0 or 1 with improvement by at least 2 grades).

#### 8.1.1 Primary Efficacy Analysis

The efficacy of the 1% OPA-15406 group will be demonstrated compared to the vehicle group based on the primary endpoint, the success rate in IGA at Week 4. The Cochran-Mantel-Haenszel test will be conducted at a two-sided significance level of 5% using the baseline IGA (2 or 3) as a stratification factor. The difference in the success rate in IGA and its two-sided 95% confidence interval (common risk difference adjusted by the Mantel-Haenszel method and its two-sided 95% confidence interval) between the vehicle group and the 1% OPA-15406 group will be determined. Also, the two-sided 95% confidence interval of the success rate in IGA in each treatment group (based on Clopper-Pearson method) will be calculated.

The SAS code for the Cochran-Mantel-Haenszel test and to determine the difference in the success rate and two-sided 95% confidence interval is as follows:

```
proc freq;
tables BaselineIGA*Treatment*Response / riskdiff(common) cmh;
run;
```

A supplementary analysis will be performed using data which includes missing data imputed by Last Observation Carried Forward (LOCF) and Observed Cases (OC) data which does not include the imputed missing data in the same manner.

Data at Weeks 1 and 2 will also be analyzed in the same manner as the primary endpoint at Week 4.

#### 8.2 Secondary Efficacy Endpoints

#### 8.2.1 Success Rates in IGA (Revised Definition) and EASI

The success rate in achieving an IGA score of 0 or 1 (revised definition from primary efficacy endpoint) by Week 4 and the success rate in EASI 75, EASI 90, and EASI 50 by Week 4 will be analyzed in the same manner as the primary endpoint in Section 8.1.1

For IGA, subjects who achieve a score of 0 or 1 in IGA will be handled as responders and subjects who do not achieve a score 0 or 1 in IGA will be handled as non-responders. Subjects with missing IGA data will be handled as non-responders.

EASI 75 will be set as the important secondary endpoint, and subjects whose percentage change in their total EASI score from baseline decreases by ≥75% will be handled as responders and subjects whose percentage change from baseline does not decrease by ≥75% will be handled as non-responders. Subjects with missing EASI 75 data will be handled as non-responders. EASI 90 and EASI 50 will be analyzed in the same manner. Similarities with the primary endpoint results will be assessed using response rates in EASI (EASI 75, EASI 90, and EASI 50).

#### 8.2.2 Change From Baseline Through Week 4 in the IGA Score

Based on the OC data set, change from baseline (Week 1, Week 2, and Week 4) will be analyzed using a mixed-model repeated measure (MMRM) with treatment (1% OPA-15406 or vehicle), timepoint, interaction between the treatment and timepoint as factors and baseline values as covariates. An unstructured covariance matrix will be used and Kenward-Roger method will be used to calculate the degree of freedom. If the MMRM procedure fails to converge under unstructured covariance structure, the

following structure will be used in the order of 1) heterogeneous toeplitz, 2) heterogeneous autoregressive of order 1, and 3) heterogeneous compound symmetry, and the first covariance structure converging will be used. The MMRM analysis with the structured error covariance matrix will use a sandwich estimator. The least square mean will be calculated by treatment group and timepoint.

The SAS code for MMRM analysis is as follows:

```
proc mixed method = reml;

class Treatment Visit Subject;

model Change = Treatment Visit Treatment*Visit Baseline / s ddfm = kr;

repeated Visit / type = un sub = Subject;

lsmeans Treatment*Visit / pdiff cl alpha = 0.05;

run;

"Baseline" is baseline IGA data. "Visit" includes data at Weeks 1, 2, and 4.

The SAS code used in the case of convergence failure is as follows: (Specify type = TOEPH for heterogeneous toeplitz, type = ARH(1) for heterogeneous autoregressive of order 1, and type = CSH for heterogeneous compound symmetry.)

proc mixed method = reml empirical;

class Treatment Visit Subject;

model Change = Treatment Visit Treatment*Visit Baseline / s;

repeated Visit / type = TOEPH sub = Subject;

lsmeans Treatment*Visit / pdiff cl alpha = 0.05;
```

Based on the OC and LOCF data sets, change from baseline at each timepoint will be analyzed using an ANCOVA model with treatment (1% OPA-15406 or vehicle) as factors and baseline IGA scores as covariates. The least square mean will be calculated at each timepoint (Weeks 1, 2, and 4) for each treatment group. Also, the difference in the least square mean between the vehicle group and the OPA-15406 group will be calculated along with its two-sided 95% confidence interval and p value. Based on the OC and LOCF data sets, the descriptive statistics will be calculated for measured values and changes from the baseline at each timepoint by treatment group.

run;

A graph will be created for the least square mean and standard deviation for the change from baseline in IGA calculated by MMRM for each treatment group.

## 8.2.3 Shift Table for Investigator's Global Assessment Scores up to Week 4

Based on the OC and LOCF data sets, a shift table will be created for IGA scores (0, 1, 2, 3, and 4) at Weeks 1, 2, and 4.

# 8.2.4 Change From Baseline Through Week 4 in the Total EASI Score and Each EASI Clinical Sign Score

Based on the OC and LOCF data sets, the analysis will be performed in the same manner as for the change from baseline in IGA scores. In addition to clinical signs (erythema, infiltration/papule, excoriation, and lichenification), scores on body regions (face, neck, and head; upper limbs; trunk; and lower limbs) will also be analyzed in the same manner. For EASI, the percentage change will also be analyzed. A graph will be created for the least square mean and standard deviation for the change from baseline in the total EASI score calculated by MMRM for each treatment group.

#### 8.2.5 Change From Baseline Through Day 8 in VRS for Pruritus

Based on the OC data set, the analysis will be performed in the same manner as for the change from baseline in IGA scores. Timepoints will include baseline through Day 8.

## 8.2.6 Change From Baseline Through Week 4 in VRS for Pruritus

Based on the OC and LOCF data sets, the analysis will be performed in the same manner as for the change from baseline in IGA scores. Timepoints will include baseline, Weeks 1, 2, and 4.

## 8.2.7 Change From Baseline Through Week 4 in the Total POEM Score

Based on the OC and LOCF data sets, the analysis will be performed in the same manner as for the change from baseline in IGA scores. The percentage change in the total POEM score will also be analyzed in the same manner.

## 8.2.8 Change From Baseline Through Week 4 in Skindex-16

Based on the OC and LOCF data sets, change from baseline in each item score, the scale score (mean score of item scores on each scale [symptoms, emotions, and functions]), and the mean score of 16 items of Skindex-16 will be analyzed in the same manner as the change from baseline in IGA scores. However, for each of the 16 items, the original 0 to

6 scale score will be converted to a 0 to 100 scale score (= original score  $\times$  100/6, rounded to 1 decimal place) for analysis.

# 8.2.9 Change From Baseline Through Week 4 in the Total Affected BSA (%)

Based on the OC and LOCF data sets, the analysis will be performed in the same manner as for the change from baseline in IGA scores.

#### 8.3 Subgroup Analyses

The success rate in IGA (IGA of 0 or 1 with improvement of at least 2 grades) and EASI 75 will be analyzed for each of the following subgroups in the same manner as the primary endpoint in Section 8.1.1.

Age: less than 30, 30 years and older

Sex: male, female

IGA score at baseline: 2 (mild), 3 (moderate)

Severity of AD: mild, moderate, severe, very severe

Total EASI score at baseline: less than 15, 15 and above

Affected BSA at baseline: less than 20%, 20% and above

## 9 Safety Analysis

The following analyses will be performed in the SS.

#### 9.1 Extent of Exposure

Based on the SS, the descriptive statistics will be presented for the total amount and the amount per dose of the IMP by treatment group and in total. Also, descriptive statistics will be presented in the same manner by taking into consideration the concentration of the IMP (1% OPA-15406 and vehicle [0%]). Where the weight of IMP at retrieval is unknown, the amount of administration will be calculated by assuming that the retrieved weight is 0.

#### 9.2 Adverse Events

All AEs will be coded by System Organ Class (SOC) and Preferred Term (PT) using the MedDRA.

For the following treatment-emergent adverse events (TEAEs) occurring after the start of IMP administration, the number and percentage of subjects will be calculated by treatment group and for all subjects. Skin and subcutaneous tissue disorders will be summarized in the same manner by grade as specified in the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 translated into Japanese by JCOG.

- TEAEs
- TEAEs resulting in death
- Serious TEAEs
- TEAEs leading to discontinuation of IMP administration
- TEAEs by severity
- TEAEs (skin and subcutaneous tissue disorders alone) by CTCAE grade
- TEAEs in treatment areas

Also, for the TEAEs and non-serious TEAEs occurring in at least 5% of subjects in each treatment group, the number and percentage of subjects will be calculated for each treatment group.

Adverse reactions (TEAEs for which a causal relationship with the IMP cannot be ruled out) will be analyzed in the same manner as TEAEs.

If the same event occurs more than once in the same subject, the most severe will be used.

#### 9.3 Clinical Laboratory Tests

For each parameter (except qualitative urinalysis), the descriptive statistics will be calculated for measured values and changes from the baseline at each timepoint by treatment group. For qualitative urinalysis values of clinical laboratory tests, a shift table at each timepoint against the baseline will be created for each treatment group. For clinical laboratory tests except qualitative urinalysis, a shift table for values before and after administration categorized as normal, high, or low relative to the reference value will be created for each treatment group.

#### 9.4 Vital Signs and Body Weight

For body weight, body temperature, blood pressure (systolic and diastolic), and pulse rate, the descriptive statistics will be calculated for measured values and changes from baseline at each timepoint by treatment group. The number and percentage of subjects with clinically abnormal changes (Appendix 1) in body temperature, blood pressure (systolic and diastolic), and pulse rate will be calculated by treatment group and for all

subjects. For clinically abnormal changes, all data after starting administration, except for baseline or missing timepoints, will be included in the evaluation. Also, a list of subjects with clinically abnormal changes will be created.

#### 9.5 Physical Examination

Not applicable.

#### 9.6 Electrocardiogram

Not applicable.

#### 9.7 Liver Function Tests

The number and percentage of subjects with abnormal changes in liver function (Appendix 2) will be calculated by treatment group. Also, a list of abnormal changes in liver function will be created. For clinically abnormal changes, all data after starting administration, except for baseline or missing timepoints, will be included in the evaluation.

## 10 Pharmacokinetic Analysis

Not applicable.

## 11 Pharmacodynamic Analysis

Not applicable.

## 12 Pharmacogenomic Analysis

Not applicable.

## 13 Interim Analysis

Not applicable.

## 14 Changes in the Planned Analyses

The following calculations specified in Section 7.6.2 in the protocol were not performed.

• The number and percentage of subjects who are in the potentially clinically significant range will be calculated.

## 15 References

None.

## **Appendix 1** Criteria for Vital Signs Potential Clinical Significance

| Variable | CRITERIA 1 | CRITERIA 2 |
|---|---|---|
| DIASTOLIC BLOOD | DIASTOLIC BLOOD PRESSURE | DIASTOLIC BLOOD PRESSURE |
| PRESSURE (mmHg) | (mmHg) <50 AND DECREASE | (mmHg) >105 AND INCREASE |
| TRESSURE (IIIIIII) | ≥15 | ≥15 |
| PULSE RATE (beats/min) | PULSE RATE (BPM) <50 AND | PULSE RATE (BPM) >120 AND |
| FOLSE KATE (beats/fillif) | DECREASE ≥15 | INCREASE ≥15 |
| SYSTOLIC BLOOD | SYSTOLIC BLOOD PRESSURE | SYSTOLIC BLOOD PRESSURE |
| PRESSURE (mmHg) | (mmHg) <90 AND DECREASE | (mmHg) >180 AND INCREASE |
| PRESSURE (IIIIIIII) | ≥20 | ≥20 |
| TEMBED ATLIBE (9C) | | TEMPERATURE (°C) ≥37.8 AND |
| TEMPERATURE (°C) | | INCREASE ≥1.1°C |
| WEIGHT (kg) | WEIGHT (kg) DECREASE ≥7% | WEIGHT (kg) INCREASE ≥7% |

## Appendix 2 Criteria for Potential Hy's Law

The potential Hy's Law Cases are defined as subjects with the following criteria: ALT>=3xULN (OR SCREENING VALUE) OR AST>=3xULN (OR SCREENING VALUE) AND BILIRUBIN>=2xULN (OR SCREENING VALUE)

## Appendix 3 List of Summary Tables

| CT-1 | Subject Disposition |
|---|---|
| CT-2 | Reasons for Discontinuation |
| CT-3.1 | Demographic Characteristics Safety Set |
| CT-3.2 | Demographic Characteristics Efficacy Set |
| CT-4.1 | Concomitant Medications: Medications Taken Prior to Start of Study<br>Therapy |
| CT-4.2 | Concomitant Medications: Medications Taken During Study Therapy |
| CT-4.3 | Concomitant Medications: Medications Taken After Study Therapy |
| CT-5.1.1 | Analysis of Responder Rate for Overall IGA Score |
| CT-5.1.2 | Supplementary Analysis of Responder Rate for Overall IGA Score - LOCF |
| CT-5.1.3 | Supplementary Analysis of Responder Rate for Overall IGA Score - OC |
| CT-5.1.4 | Analysis of Responder Rate for Overall IGA Score - Revised Responder Definition |
| CT-5.1.5 | Shift Tables of Overall IGA Score - OC |
| CT-5.1.6 | Shift Tables of Overall IGA Score - LOCF |
| CT-5.2.1 | Analysis of 75% Over Responder Rate for Overall EASI Score |
| CT-5.2.2 | Analysis of 90% Over Responder Rate for Overall EASI Score |
| CT-5.2.3 | Analysis of 50% Over Responder Rate for Overall EASI Score |
| CT-5.3.1 | Analysis of Baseline and Change from Baseline in Overall IGA Score - MMRM |
| CT-5.3.2 | Analysis of Baseline and Change from Baseline in Overall IGA Score - ANCOVA OC |
| CT-5.3.3 | Analysis of Baseline and Change from Baseline in Overall IGA Score - ANCOVA LOCF |
| CT-5.4.1.1 | Analysis of Baseline and Change from Baseline in Overall EASI Score - MMRM |

| CT-5.4.1.2 | Analysis of Baseline and Change from Baseline in Overall EASI Score - ANCOVA OC |
|---|---|
| CT-5.4.1.3 | Analysis of Baseline and Change from Baseline in Overall EASI Score - ANCOVA LOCF |
| CT-5.4.1.4 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score - MMRM |
| CT-5.4.1.5 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score - ANCOVA OC |
| CT-5.4.1.6 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score - ANCOVA LOCF |
| CT-5.4.2.1 | Analysis of Baseline and Change from Baseline in Overall EASI Score, Erythema - MMRM |
| CT-5.4.2.2 | Analysis of Baseline and Change from Baseline in Overall EASI Score, Erythema - ANCOVA OC |
| CT-5.4.2.3 | Analysis of Baseline and Change from Baseline in Overall EASI Score, Erythema - ANCOVA LOCF |
| CT-5.4.2.4 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Erythema - MMRM |
| CT-5.4.2.5 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Erythema - ANCOVA OC |
| CT-5.4.2.6 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Erythema - ANCOVA LOCF |
| CT-5.4.3.1 | Analysis of Baseline and Change from Baseline in Overall EASI Score, Induration/Papulation - MMRM |
| CT-5.4.3.2 | Analysis of Baseline and Change from Baseline in Overall EASI Score, Induration/Papulation - ANCOVA OC |
| CT-5.4.3.3 | Analysis of Baseline and Change from Baseline in Overall EASI Score, Induration/Papulation - ANCOVA LOCF |
| CT-5.4.3.4 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Induration/Papulation - MMRM |
| CT-5.4.3.5 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Induration/Papulation - ANCOVA OC |

| CT-5.4.3.6 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Induration/Papulation - ANCOVA LOCF |
|---|---|
| CT-5.4.4.1 | Analysis of Baseline and Change from Baseline in Overall EASI Score, Excoriation - MMRM |
| CT-5.4.4.2 | Analysis of Baseline and Change from Baseline in Overall EASI Score, Excoriation - ANCOVA OC |
| CT-5.4.4.3 | Analysis of Baseline and Change from Baseline in Overall EASI Score, Excoriation - ANCOVA LOCF |
| CT-5.4.4.4 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Excoriation - MMRM |
| CT-5.4.4.5 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Excoriation - ANCOVA OC |
| CT-5.4.4.6 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Excoriation - ANCOVA LOCF |
| CT-5.4.5.1 | Analysis of Baseline and Change from Baseline in Overall EASI Score,<br>Lichenification - MMRM |
| CT-5.4.5.2 | Analysis of Baseline and Change from Baseline in Overall EASI Score,<br>Lichenification - ANCOVA OC |
| CT-5.4.5.3 | Analysis of Baseline and Change from Baseline in Overall EASI Score,<br>Lichenification - ANCOVA LOCF |
| CT-5.4.5.4 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Lichenification - MMRM |
| CT-5.4.5.5 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Lichenification - ANCOVA OC |
| CT-5.4.5.6 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Lichenification - ANCOVA LOCF |
| CT-5.4.6.1 | Analysis of Baseline and Change from Baseline in Overall EASI Score, HEAD/NECK - MMRM |
| CT-5.4.6.2 | Analysis of Baseline and Change from Baseline in Overall EASI Score, HEAD/NECK - ANCOVA OC |
| CT-5.4.6.3 | Analysis of Baseline and Change from Baseline in Overall EASI Score, |

| CT-5.4.6.4 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, HEAD/NECK - MMRM |
|---|---|
| CT-5.4.6.5 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, HEAD/NECK - ANCOVA OC |
| CT-5.4.6.6 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, HEAD/NECK - ANCOVA LOCF |
| CT-5.4.7.1 | Analysis of Baseline and Change from Baseline in Overall EASI Score, UPPER LIMBS - MMRM |
| CT-5.4.7.2 | Analysis of Baseline and Change from Baseline in Overall EASI Score, UPPER LIMBS - ANCOVA OC |
| CT-5.4.7.3 | Analysis of Baseline and Change from Baseline in Overall EASI Score, UPPER LIMBS - ANCOVA LOCF |
| CT-5.4.7.4 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, UPPER LIMBS - MMRM |
| CT-5.4.7.5 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, UPPER LIMBS - ANCOVA OC |
| CT-5.4.7.6 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, UPPER LIMBS - ANCOVA LOCF |
| CT-5.4.8.1 | Analysis of Baseline and Change from Baseline in Overall EASI Score, TRUNK - MMRM |
| CT-5.4.8.2 | Analysis of Baseline and Change from Baseline in Overall EASI Score, TRUNK - ANCOVA OC |
| CT-5.4.8.3 | Analysis of Baseline and Change from Baseline in Overall EASI Score, TRUNK - ANCOVA LOCF |
| CT-5.4.8.4 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, TRUNK - MMRM |
| CT-5.4.8.5 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, TRUNK - ANCOVA OC |
| CT-5.4.8.6 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, TRUNK - ANCOVA LOCF |
| CT-5.4.9.1 | Analysis of Baseline and Change from Baseline in Overall EASI Score, LOWER LIMBS - MMRM |

| CT-5.4.9.2 | Analysis of Baseline and Change from Baseline in Overall EASI Score, LOWER LIMBS - ANCOVA OC |
|---|---|
| CT-5.4.9.3 | Analysis of Baseline and Change from Baseline in Overall EASI Score, LOWER LIMBS - ANCOVA LOCF |
| CT-5.4.9.4 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, LOWER LIMBS - MMRM |
| CT-5.4.9.5 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, LOWER LIMBS - ANCOVA OC |
| CT-5.4.9.6 | Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, LOWER LIMBS - ANCOVA LOCF |
| CT-5.5.1 | Analysis of Baseline and Change from Baseline in VRS for Pruritus Score - MMRM |
| CT-5.5.2 | Analysis of Baseline and Change from Baseline in VRS for Pruritus Score - ANCOVA OC |
| CT-5.5.3 | Analysis of Baseline and Change from Baseline in VRS for Pruritus Score - ANCOVA LOCF |
| CT-5.5.4 | Analysis of Baseline and Change from Baseline in VRS for Pruritus Score (Week 1) - MMRM |
| CT-5.5.5 | Analysis of Baseline and Change from Baseline in VRS for Pruritus Score (Week 1) - ANCOVA OC |
| CT-5.6.1 | Analysis of Baseline and Change from Baseline in POEM Score - MMRM |
| CT-5.6.2 | Analysis of Baseline and Change from Baseline in POEM Score - ANCOVA OC |
| CT-5.6.3 | Analysis of Baseline and Change from Baseline in POEM Score - ANCOVA LOCF |
| CT-5.6.4 | Analysis of Baseline and Percent Change from Baseline in POEM Score - MMRM |
| CT-5.6.5 | Analysis of Baseline and Percent Change from Baseline in POEM Score - ANCOVA OC |
| CT-5.6.6 | Analysis of Baseline and Percent Change from Baseline in POEM Score - ANCOVA LOCF |

| CT-5.7.1.1 | Analysis of Baseline and Change from Baseline in Skindex-16 - MMRM |
|---|---|
| CT-5.7.1.2 | Analysis of Baseline and Change from Baseline in Skindex-16 - ANCOVA OC |
| CT-5.7.1.3 | Analysis of Baseline and Change from Baseline in Skindex-16 - ANCOVA LOCF |
| CT-5.7.2.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Symptoms - MMRM |
| CT-5.7.2.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Symptoms - ANCOVA OC |
| CT-5.7.2.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Symptoms - ANCOVA LOCF |
| CT-5.7.3.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Emotions - MMRM |
| CT-5.7.3.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Emotions - ANCOVA OC |
| CT-5.7.3.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Emotions - ANCOVA LOCF |
| CT-5.7.4.1 | Analysis of Baseline and Change from Baseline in Skindex-16,<br>Functioning - MMRM |
| CT-5.7.4.2 | Analysis of Baseline and Change from Baseline in Skindex-16,<br>Functioning - ANCOVA OC |
| CT-5.7.4.3 | Analysis of Baseline and Change from Baseline in Skindex-16,<br>Functioning - ANCOVA LOCF |
| CT-5.7.5.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 1 - MMRM |
| CT-5.7.5.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 1 - ANCOVA OC |
| CT-5.7.5.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 1 - ANCOVA LOCF |
| CT-5.7.6.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 2 - MMRM |

| CT-5.7.6.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 2 - ANCOVA OC |
|---|---|
| CT-5.7.6.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 2 - ANCOVA LOCF |
| CT-5.7.7.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 3 - MMRM |
| CT-5.7.7.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 3 - ANCOVA OC |
| CT-5.7.7.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 3 - ANCOVA LOCF |
| CT-5.7.8.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 4 - MMRM |
| CT-5.7.8.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 4 - ANCOVA OC |
| CT-5.7.8.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 4 - ANCOVA LOCF |
| CT-5.7.9.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 5 - MMRM |
| CT-5.7.9.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 5 - ANCOVA OC |
| CT-5.7.9.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 5 - ANCOVA LOCF |
| CT-5.7.10.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 6 - MMRM |
| CT-5.7.10.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 6 - ANCOVA OC |
| CT-5.7.10.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 6 - ANCOVA LOCF |
| CT-5.7.11.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 7 - MMRM |
| CT-5.7.11.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 7 - ANCOVA OC |

| CT-5.7.11.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 7 - ANCOVA LOCF |
|---|---|
| CT-5.7.12.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 8 - MMRM |
| CT-5.7.12.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 8 - ANCOVA OC |
| CT-5.7.12.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 8 - ANCOVA LOCF |
| CT-5.7.13.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 9 - MMRM |
| CT-5.7.13.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 9 - ANCOVA OC |
| CT-5.7.13.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 9 - ANCOVA LOCF |
| CT-5.7.14.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 10 MMRM |
| CT-5.7.14.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 10 ANCOVA OC |
| CT-5.7.14.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 10 ANCOVA LOCF |
| CT-5.7.15.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 11 MMRM |
| CT-5.7.15.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 11 ANCOVA OC |
| CT-5.7.15.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 11 ANCOVA LOCF |
| CT-5.7.16.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 12 MMRM |
| CT-5.7.16.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 12 ANCOVA OC |

ANCOVA LOCF

CT-5.7.16.3

Analysis of Baseline and Change from Baseline in Skindex-16, Item 12 -

| CT-5.7.17.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 13 - MMRM |
|---|---|
| CT-5.7.17.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 13 - ANCOVA OC |
| CT-5.7.17.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 13 - ANCOVA LOCF |
| CT-5.7.18.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 14 - MMRM |
| CT-5.7.18.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 14 - ANCOVA OC |
| CT-5.7.18.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 14 - ANCOVA LOCF |
| CT-5.7.19.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 15 - MMRM |
| CT-5.7.19.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 15 - ANCOVA OC |
| CT-5.7.19.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 15 - ANCOVA LOCF |
| CT-5.7.20.1 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 16 - MMRM |
| CT-5.7.20.2 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 16 - ANCOVA OC |
| CT-5.7.20.3 | Analysis of Baseline and Change from Baseline in Skindex-16, Item 16 - ANCOVA LOCF |
| CT-5.8.1 | Analysis of Baseline and Change from Baseline in Overall Percentage<br>Affected Body Surface Area - MMRM |
| CT-5.8.2 | Analysis of Baseline and Change from Baseline in Overall Percentage<br>Affected Body Surface Area - ANCOVA OC |
| CT-5.8.3 | Analysis of Baseline and Change from Baseline in Overall Percentage<br>Affected Body Surface Area - ANCOVA LOCF |
| CT-6.1.1 | Subgroup Analysis of Responder Rate for Overall IGA Score - by Age |

| CT-6.1.2 | Subgroup Analysis of Responder Rate for Overall IGA Score - by Sex |
|---|---|
| CT-6.1.3 | Subgroup Analysis of Responder Rate for Overall IGA Score - by IGA Score at Baseline |
| CT-6.1.4 | Subgroup Analysis of Responder Rate for Overall IGA Score - by Severity of Atopic Dermatitis |
| CT-6.1.5 | Subgroup Analysis of Responder Rate for Overall IGA Score - by Total EASI Score at Baseline (<15, 15=<) |
| CT-6.1.6 | Subgroup Analysis of Responder Rate for Overall IGA Score - by Affected Body Surface Area (<20%, 20%=<) |
| CT-6.2.1 | Subgroup Analysis of 75% Over Responder Rate for Overall EASI Score by Age |
| CT-6.2.2 | Subgroup Analysis of 75% Over Responder Rate for Overall EASI Score by Sex |
| CT-6.2.3 | Subgroup Analysis of 75% Over Responder Rate for Overall EASI Score by IGA Score at Baseline |
| CT-6.2.4 | Subgroup Analysis of 75% Over Responder Rate for Overall EASI Score by Severity of Atopic Dermatitis |
| CT-6.2.5 | Subgroup Analysis of 75% Over Responder Rate for Overall EASI Score - by Total EASI Score at Baseline (<15, 15=<) |
| CT-6.2.6 | Subgroup Analysis of 75% Over Responder Rate for Overall EASI Score by Affected Body Surface Area (<20%, 20%=<) |
| CT-7.1.1 | Summary of Treatment Compliance |
| CT-7.1.2 | Summary of Treatment Compliance for Number of Administrations |
| CT-7.2.1 | Extent of Exposure to Trial Medication |
| CT-7.2.2 | Summary of Exposure to Trial Medication |
| CT-8.1.1 | Adverse Events (All Causalities) |
| CT-8.1.2 | Adverse Events According to Application Site (All Causalities) |
| CT-8.2.1 | Incidence of Treatment-emergent Adverse Events by System Organ Class |
| CT-8.2.2 | Incidence of Treatment-emergent Adverse Events by System Organ Class and Preferred Term |

| CT-8.2.3 | Incidence of Treatment-emergent Adverse Events by System Organ Class,<br>Preferred Term and Severity |
|---|---|
| CT-8.2.4 | Incidence of Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade |
| CT-8.3.1 | Incidence of Potentially Drug-Related Treatment-emergent Adverse<br>Events by System Organ Class |
| CT-8.3.2 | Incidence of Potentially Drug-Related Treatment-emergent Adverse<br>Events by System Organ Class and Preferred Term |
| CT-8.3.3 | Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity |
| CT-8.3.4 | Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade |
| CT-8.4.1 | Incidence of Deaths due to Treatment-emergent Adverse Events by<br>System Organ Class |
| CT-8.4.2 | Incidence of Deaths due to Treatment-emergent Adverse Events by<br>System Organ Class and Preferred Term |
| CT-8.5.1 | Incidence of Serious Treatment-emergent Adverse Events by System<br>Organ Class |
| CT-8.5.2 | Incidence of Serious Treatment-emergent Adverse Events by System<br>Organ Class and Preferred Term |
| CT-8.5.3 | Incidence of Serious Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity |
| CT-8.5.4 | Incidence of Serious Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade |
| CT-8.6.1 | Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class |
| CT-8.6.2 | Incidence of Treatment-emergent Adverse Events Resulting in<br>Discontinuation from Study by System Organ Class and Preferred Term |
| CT-8.6.3 | Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class, Preferred Term and Severity |

| CT-8.6.4 | Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class, Preferred Term and CTCAE Grade |
|---|---|
| CT-8.7 | Incidence of Treatment-emergent Adverse Events Greater Than or Equal to 5% in Any Group by System Organ Class and Preferred Term |
| CT-8.8 | Incidence of Non-Serious Treatment-emergent Adverse Events Greater<br>Than or Equal to 5% in Any Group by System Organ Class and Preferred<br>Term |
| CT-8.9 | Incidence of Treatment-emergent Adverse Events by System Organ Class and Preferred Term According to Application Site |
| CT-8.10 | Incidence of Potentially Drug-related Treatment-emergent Adverse Events<br>by System Organ Class and Preferred Term According to Application Site |
| CT-9.1 | Listing of Deaths |
| CT-9.2 | Listing of Serious Adverse Events |
| CT-9.3 | Listing of Study Drug Discontinuations Due to Adverse Events |
| CT-9.4 | Incidence of Potential Hy's Law Cases |
| CT-9.5 | Listing of Potential Hy's Law Cases - by Subject |
| CT-10.1.1 | Mean Change From Baseline in Laboratory Test Values: Serum Chemistry |
| CT-10.1.2 | Mean Change From Baseline in Laboratory Test Values: Hematology |
| CT-10.2.1 | Shift Tables of Clinical Laboratory Test Results: Serum Chemistry |
| CT-10.2.2 | Shift Tables of Clinical Laboratory Test Results: Hematology |
| CT-10.2.3 | Shift Tables of Clinical Laboratory Test Results: Urinalysis |
| CT-11.1 | Mean Change From Baseline in Vital Sign Parameters |
| CT-11.2 | Listing of Vital Signs Abnormalities |
| CT-11.3 | Incidence of Potential Clinical Significance in Vital Signs |
| CT-11.4 | Criteria for Vital Signs Potential Clinical Significance |
| CF-1.1 | Incidence of Responder Rate for Overall IGA Score by Visit |
| CF-1.2 | Incidence of 75% Over Responder Rate for Overall EASI Score by Visit |

#### Protocol 271-102-00007

| CF-1.3 | Incidence of 90% Over Responder Rate for Overall EASI Score by Visit |
|---|---|
| CF-1.4 | Incidence of 50% Over Responder Rate for Overall EASI Score by Visit |
| CF-2.1 | Least Square Means of Change from Baseline in Overall IGA Score by Visit - MMRM |
| CF-2.2 | Least Square Means of Change from Baseline in Overall EASI Score by Visit - MMRM |

## **Appendix 4** List of Subject Data Listings

| PDATA-1.1 | Inclusion and Exclusion Criteria Not Met |
|---|---|
| PDATA-1.2 | Subject Disposition |
| PDATA-2.1 | Medical History |
| PDATA-2.2 | History of Atopic Dermatitis |
| PDATA-3.1 | Concomitant Medications and Therapy Taken Prior to Start of Study<br>Therapy |
| PDATA-3.2 | Concomitant Medications and Therapy Taken During Study Therapy |
| PDATA-3.3 | Concomitant Medications and Therapy Taken After Study Therapy |
| PDATA-4.1 | Exposure to Trial Medication |
| PDATA-4.2 | Listing of Trial Medication by Subject |
| PDATA-5.1 | Physical Examination |
| PDATA-6 | Adverse Events |
| PDATA-7 | Vital Signs |
| PDATA-8 | Screening Failures |
| PDATA-9 | Protocol Deviations (Major) - CRF |
| PDATA-10 | Patch Application and Removal |
| PDATA-11 | Overall Investigator's Global Assessment of Disease Severity |
| PDATA-12 | Eczema Area and Severity Index |
| PDATA-13 | Verbal Rating Scale |
| PDATA-14 | Patient-Oriented Eczema Measure |
| PDATA-15 | Affected Body Surface Area |
| PDATA-16 | Treatment Area |
| PDATA-17 | Skindex-16 Score |

| DEMOG-1 | Demographic Characteristics |
|---|---|
| DEMOG-2 | Informed Consent |
| AE-1 | Adverse Events |
| SMED-1 | Investigational Medicinal Product Compliance |
| SMED-2 | Actual Exposure to Study Medication |
| SMED-3 | Investigational Medicinal Product Compliance for Number of<br>Administrations |
| EFF-1 | Change from Baseline in IGA Score and Response with Overall IGA Score |
| EFF-2 | Change from Baseline in Total EASI Score |
| EFF-3 | Change from Baseline in EASI Score, Erythema |
| EFF-4 | Change from Baseline in EASI Score, Induration/Papulation |
| EFF-5 | Change from Baseline in EASI Score, Excoriation |
| EFF-6 | Change from Baseline in EASI Score, Lichenification |
| EFF-7 | Change from Baseline in EASI Score, HEAD/NECK |
| EFF-8 | Change from Baseline in EASI Score, UPPER LIMBS |
| EFF-9 | Change from Baseline in EASI Score, TRUNK |
| EFF-10 | Change from Baseline in EASI Score, LOWER LIMBS |
| EFF-11 | Change from Baseline in VRS Score |
| EFF-12 | Change from Baseline in POEM Score |
| EFF-13 | Change from Baseline in Overall Percentage Affected Body Surface Area |
| EFF-14 | Change from Baseline in Skindex-16 Score, Skindex-16 Average Scale |
| EFF-15 | Change from Baseline in Skindex-16 Score, Symptoms Average Scale |
| EFF-16 | Change from Baseline in Skindex-16 Score, Emotions Average Scale |

#### Protocol 271-102-00007

| EFF-17 | Change from Baseline in Skindex-16 Score, Functioning Average Scale |
|---|---|
| LAB-1 | Laboratory Test Results: Serum Chemistry |
| LAB-2 | Laboratory Test Results: Hematology |
| LAB-3 | Laboratory Test Results: Urinalysis |
| PDEV-1 | Summary of Subjects with Major Protocol Deviations by Type of Deviation |
| SUBEX-1 | Subjects Excluded From Analysis Set |